CLINICAL TRIAL: NCT02700178
Title: Development of a Biofeedback Intervention to Reduce the Risk of Upper Extremity Overuse Injury Following Paraplegia and Tetraplegia
Brief Title: Biofeedback for Wheelchair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kristin Zhao, PhD, Director, Assistive and Restorative Technology Laboratory, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-008240
Record Dates: First submitted 2016-02-17; First posted 2016-03-07 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biofeedback (Experimental): Participants will be asked to participate in all or a subset of daily activities for wheelchair users. The intervention will consist of visual and/or auditory cues to guide their movement while performing the tasks during one to two sessions.
  Interventions: Other: Biofeedback

INTERVENTIONS:
Other: Biofeedback — The visual biofeedback will consist of line or shape targets on a screen that the participants will aim to achieve with your movements. The auditory cues will be a tone or multiple tones to alert them when to move and/or when targets have been achieved. During the biofeedback session the study staff may also provide verbal cues and feedback.

SUMMARY:
This study will evaluate movement of the arm and forces put through the hand during activities performed in a manual wheelchair. The goal of this study is to identify what motions and forces are most likely to lead to the development of pain or pathology and determine the feasibility of strategies to modify movements and decrease risk.

DETAILED DESCRIPTION:
Participants in the study will be asked to participate in the following during the first (1st) session:

1. Physical exam assessing joint motion
2. Questionnaires asking about shoulder pain
3. All or a subset of the following activities:

   1. Level wheelchair propulsion for up to 10 minutes
   2. Ramp wheelchair propulsion
   3. Lifting the wheelchair, including into a car (simulated car in therapy area)
   4. Transferring in/out of the wheelchair
   5. Overhead tasks (such as lifting an object off a shelf)
   6. Reaching

During the next session(s), participants will be asked to participate in all or a subset of the activities listed above (3a-3f) and will also be guided through a biofeedback intervention. The intervention will consist of visual and/or auditory cues to guide movement while performing the tasks. The visual biofeedback will consist of line or shape targets on a screen that are the participant's goal to achieve with their movements. The auditory cues will be a tone or multiple tones to alert the participant when to move and/or when targets have been achieved. During the biofeedback session the study staff may also provide verbal cues and feedback.

The investigators may review the medical records of the participants to obtain information about their spinal cord injury, wheelchair and any injury to their muscles, ligaments, bones or nerves.

During all sessions, and prior to performing the activities listed (3a-3f), motion sensors will be applied to the skin overlying the participant's sternum (chest), shoulder blade, via a plastic cuff on the arm just above the elbow, and wrist using medical grade adhesive tape. Sensors that detect muscle activity may also be applied to the skin of the participant's arm. Sensors that detect force applied by the participant's arm will also be used.

Force will be detected using all or a subset of the following tools: exchanging one of the wheels on the participant's wheelchair for one of the same size that detects force, having the participant wear a glove that detects force, and using a mat that detects force.

The activities completed while in this study may be photographed or videotaped.

ELIGIBILITY:
Individuals with spinal cord injury (paraplegia and tetraplegia)

Inclusion Criteria:

1. Age 18-60 at time of enrollment
2. Spinal cord injury or disease leading to paraplegia or tetraplegia
3. Uses a manual wheelchair as primary mode of mobility
4. Independently mobile enough to participate in the study
5. Active shoulder and wrist range of motion within limits needed for the tasks performed during the study

Exclusion Criteria:

1. Surgery or significant injury to the shoulder(s) or wrist(s) of interest (such as dislocation, fracture or full rotator cuff tear) in which return to pre-injury functional status was NOT attained
2. Peripheral nerve impairment of the upper extremity being tested
3. Evidence of significant denervation of multiple scapular muscles
4. Shoulder or wrist instability on the upper extremity to be tested
5. Allergy to medical grade adhesive tape (used to secure sensors to skin)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
change in risk of shoulder impingement | approximately 6 months
  Risk of shoulder impingement, based on the relative orientation of the humerus and scapula during activities of daily living, will be evaluated at the first appointment and following the biofeedback intervention. The change in this outcome will be evaluated for significance.

SECONDARY OUTCOMES:
change in wrist posture | approximately 6 months
  Wrist posture, the position of the hand relative to the forearm, during high levels of loading will be evaluated at the first appointment and following the biofeedback intervention. The change in this outcome will be evaluated for significance.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Zhao, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials